CLINICAL TRIAL: NCT05115045
Title: Plasma SARS-CoV-2 RNA Levels in Critically Ill COVID-19 Patients (pRNA-COVID-ICU)
Brief Title: Plasma SARS-CoV-2 RNA Levels in Critically Ill COVID-19 Patients
Acronym: pRNA-COVID-ICU
Status: Completed | Type: Observational
Sponsor: Hopital of Melun (Other)
Responsible Party: Principal Investigator, Sebastien Jochmans, MD, Head of Clinical Research Unit, Hopital of Melun
Other Study IDs: 2021-MIR-05
Record Dates: First submitted 2021-11-09; First posted 2021-11-10 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Pneumonia; ARDS Due to Disease Caused by Severe Acute Respiratory Syndrome Coronavirus 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: plasmatic SARS-CoV-2 RNA quantification — plasmatic SARS-CoV-2 RNA was quantified by droplet digital PCR

SUMMARY:
Retrospective, observationnal study. Evaluation of the association between plasmatic SARS-CoV-2 RNA and day 60 mortality in ICU adult COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* in ICU hospitalization
* COVID-19 related pneumonia confirmed by PCR

Exclusion Criteria:

* plasmatic SARS-COV-2 RNA quantification not available
* patient's refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the 34 bed ICU of the Melun-Senart Hospital between march 2021 4th and june 2021 24th meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Day 60 mortality | 60 days
  Association between plasmatic SARS-CoV-2 RNA level and mortality

CONTACTS AND LOCATIONS:
Overall Officials: SEBASTIEN JOCHMANS, Study Director — GHSIF MELUN
Locations (1):
- Groupe Hospitalier Sud Ile de France, Hôpital de Melun-Sénart, Melun, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Veyer D, Kerneis S, Poulet G, Wack M, Robillard N, Taly V, L'Honneur AS, Rozenberg F, Laurent-Puig P, Belec L, Hadjadj J, Terrier B, Pere H. Highly Sensitive Quantification of Plasma Severe Acute Respiratory Syndrome Coronavirus 2 RNA Sheds Light on its Potential Clinical Value. Clin Infect Dis. 2021 Nov 2;73(9):e2890-e2897. doi: 10.1093/cid/ciaa1196. PMID 32803231